CLINICAL TRIAL: NCT05388214
Title: An Exercise and COgnitive Rehabilitation Intervention for Older Cancer Survivors (The E-Co Study)
Brief Title: Exercise and Cognitive Rehab in Older Cancer Survivors
Acronym: E-Co
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Not currently enrolling subjects.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC22022
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: geriatric oncology, cancer survivors, exercise, cognitive rehabilitation, cognition
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Memory and Attention Adaptation Training-Geriatrics (MAAT-G) is a cognitive behavioral therapy-based cognitive rehab intervention developed to address CRCD in older adults with cancer and is delivered over the course of 10 individual workshops with a trained health professional. MAAT-G focuses on an individual's psychological response to injury as compared to the biological events triggering cognitive dysfunction, and provides education and training in adaptive behavioral coping skills, stress management techniques, and compensation strategies. Geriatric Oncology-Exercise for Cancer Patients (GO-EXCAP) leverages a mobile app to deliver an individually tailored, low-to-moderate intensity, home-based walking and progressive resistance exercise program designed for patients with cancer, tailored to their physical capacity. The E-Co intervention will integrate components of GO-EXCAP into MAAT-G.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-Co (Experimental): The E-Co intervention will integrate active components of a mobile health exercise intervention (GO-EXCAP) into a cognitive rehabilitation intervention (MAAT-G).
  Interventions: Behavioral: E-Co

INTERVENTIONS:
Behavioral: E-Co — The E-Co intervention will integrate active components of a mobile health exercise intervention (GO-EXCAP) into a cognitive rehabilitation intervention (MAAT-G).

SUMMARY:
The objective of the study is to evaluate the feasibility of a combined mobile health exercise and cognitive rehabilitation intervention and its effect on cognition in a single-arm pilot study that recruits cancer survivors.

DETAILED DESCRIPTION:
Cancer survivors (i.e., those who completed cancer-directed treatment) often experience long-term treatment-related effects, such as cancer-related cognitive decline (CRCD). Exercise and cognitive rehabilitation (rehab) interventions have been shown to improve CRCD symptoms in both cancer and non-cancer populations. Among older adults without cancer, studies have also demonstrated that multicomponent interventions combining exercise and cognitive rehab are more effective in improving cognitive dysfunction than either intervention alone. However, exercise adherence and self-efficacy are lower in older adults compared to younger adults, and combined interventions may be too demanding for older cancer survivors. Therefore, innovative ways are needed to integrate an exercise program within the context of a cognitive rehab program to increase exercise adherence and self-efficacy, and ultimately improve CRCD symptoms through a streamlined multicomponent intervention.

In this study, the investigators propose to refine a multicomponent Exercise and COgnitive rehab intervention (E-Co) and assess its feasibility in older cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years at the time of consent
* Have a diagnosis of any cancer
* Have completed curative intent treatments

  * Patients on endocrine therapies are allowed to enroll
  * Patients with hematologic malignancies after autologous or allogeneic stem cell transplant are allowed to enroll as long as they have completed curative-intent treatment
* Have concerns about memory or other thinking abilities following cancer treatment*
* English speaking (because the interventions are available in English language only)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* No medical contraindications for exercise per oncologist#
* Able to walk 4 meters#
* Able to provide informed consent#

(*) Confirmed by asking the patient (#) Confirmed through eligibility confirmation with the patient's oncologist or their designee

Exclusion Criteria:

* Physical, psychological, or social impairments that would interfere with patient's ability to participate in the study or participate in the intervention, as determined by the PIs and oncology team.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Post-intervention at week 12
  Feasibility is defined based on adherence to the intervention components: 1) At least 70% of patients provide exercise data on 50% on the intervention days; and 2) At least 70% of patients attend at least 8/10 of the MAAT-G workshops.

SECONDARY OUTCOMES:
Self-reported cognition | Baseline and post-intervention at week 12
  Functional Assessment of Cancer Therapy-Cognition (FACT-Cog): The FACT-Cog is a validated patient reported outcome measure created to assess cognitive challenges identified by patients with cancer. It has 37 items and has four domains in Perceived Cognitive Impairments (PCI), Impact of PCI on Quality of Life, Comments from Others, and Perceived Cognitive Abilities. Score ranges from 0-148, higher score indicates better self-reported cognition.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline and post-intervention at week 12
  The CANTAB Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory, for non-verbalisable patterns. The subject is shown a complex visual pattern, followed by four similar patterns after a brief delay. The subject must select the pattern which exactly matches the sample. Better speed of response and higher number of correct patterns indicate better health outcomes. (Patients only)
Controlled Oral Word Association (COWA) | Baseline and post-intervention at week 12
  The Controlled Oral Word Association (COWA) tool is a measure of verbal fluency evaluating expressive language and executive function. Subjects are asked to freely generate as many words as they can that start with one of the prompted letters ("C", "F", and "L") in the span of one minute. Greater numbers of words indicate better health outcomes.
Hopkins Verbal Learning Test-Revised (HVLT-R) | Baseline and post-intervention at week 12
  The Hopkins Verbal Learning Test-Revised (HVLT-R) tool is a test of verbal learning and memory. Researchers read a list of 12 words to subjects and ask them to report as many of the words as they can recall. The reporting period is timed. Higher numbers of correctly remembered words, along with lower reporting times, are indicative of better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators if requested. Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years after study completion